CLINICAL TRIAL: NCT04099264
Title: Effect of Personalized Musical Intervention on Burden of Care in Dental Implant Surgery: A Pilot Randomized Controlled Trial
Brief Title: Effect of Music on Burden of Dental Implant Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Nathalie Gosselin, PhD, Neuropsychologist, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 18-004-CERC-P
Record Dates: First submitted 2018-08-24; First posted 2019-09-23 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Personalized Musical Intervention
Keywords: personalized musical intervention; experimental study; dissatisfaction; anxiety; surgical pain; burden of care; pilot randomized controlled trial
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Personalized music (Experimental): This arm will receive an intervention which will be personalized music. It will be provided by Music Care application (https://www.music-care.com/fr).
  Interventions: Other: Personalized music
- Control: Audio Books (Active Comparator): Control will consist of audio books.
  Interventions: Other: Audio Books

INTERVENTIONS:
Other: Personalized music — Patients in the intervention group will listen to personalized music from the Musicare application
  Arms: Intervention group: Personalized music
Other: Audio Books — Patients in the active comparator group will listen to audio books
  Arms: Control: Audio Books

SUMMARY:
Personnalized music can decrease the burden of care.

This experimental clinical trial examines the effect of personalized musical intervention on the burden of dental implant surgery. The intervention consists of a personnalized musical intervention and the control group consists of audio books. The burden of dental implant surgery will be defined by a composite variable including surgical pain, state anxiety and dissatisfaction with dental implant surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients included in the study:

* will have an adequate understanding of the French or English language both written and spoken,
* will have the physical and psychological ability to understand and complete the questionnaires used in the study,
* will consent to follow research instructions,
* will consent to follow the allocated sequence of interventions without prior notification,
* will undergo a dental implant surgery not exceeding 2 hours,

Exclusion Criteria:

Patients :

* do not have the necessary clinical criteria to receive implants.
* have an implant surgical treatment that would increase treatment time beyond 2 hours,
* have a history of neurological disorders, diagnosed with severe psychiatric disorders (e.g. schizophrenia, bipolar disorder), substance abuse
* have a major diagnosed hearing problem.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Burden of dental implant surgery | Measured immediately at the end of surgery
  Composite outcome by summing the means of the 0-10 visual analogue scales of surgical pain, state anxiety and dissatisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Gosselin, PhD, Principal Investigator — Université de Montréal, MUSEC
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bradt J, Teague A. Music interventions for dental anxiety. Oral Dis. 2018 Apr;24(3):300-306. doi: 10.1111/odi.12615. Epub 2017 Jan 5. PMID 27886431
- [Result] Carter AE, Carter G, Boschen M, AlShwaimi E, George R. Pathways of fear and anxiety in dentistry: A review. World J Clin Cases. 2014 Nov 16;2(11):642-53. doi: 10.12998/wjcc.v2.i11.642. PMID 25405187
- [Result] Cohen SM, Fiske J, Newton JT. The impact of dental anxiety on daily living. Br Dent J. 2000 Oct 14;189(7):385-90. doi: 10.1038/sj.bdj.4800777. PMID 11081950
- [Result] Gordon D, Heimberg RG, Tellez M, Ismail AI. A critical review of approaches to the treatment of dental anxiety in adults. J Anxiety Disord. 2013 May;27(4):365-78. doi: 10.1016/j.janxdis.2013.04.002. Epub 2013 Apr 13. PMID 23746494
- [Result] Hole J, Hirsch M, Ball E, Meads C. Music as an aid for postoperative recovery in adults: a systematic review and meta-analysis. Lancet. 2015 Oct 24;386(10004):1659-71. doi: 10.1016/S0140-6736(15)60169-6. Epub 2015 Aug 12. PMID 26277246
- [Result] Kuhlmann AYR, de Rooij A, Kroese LF, van Dijk M, Hunink MGM, Jeekel J. Meta-analysis evaluating music interventions for anxiety and pain in surgery. Br J Surg. 2018 Jun;105(7):773-783. doi: 10.1002/bjs.10853. Epub 2018 Apr 17. PMID 29665028
- [Result] Mejia-Rubalcava C, Alanis-Tavira J, Mendieta-Zeron H, Sanchez-Perez L. Changes induced by music therapy to physiologic parameters in patients with dental anxiety. Complement Ther Clin Pract. 2015 Nov;21(4):282-6. doi: 10.1016/j.ctcp.2015.10.005. Epub 2015 Oct 27. PMID 26573456
- [Result] Rainville P, Bao QVH, Chretien P. Pain-related emotions modulate experimental pain perception and autonomic responses. Pain. 2005 Dec 5;118(3):306-318. doi: 10.1016/j.pain.2005.08.022. Epub 2005 Nov 14. PMID 16289802
- [Result] Roy M, Peretz I, Rainville P. Emotional valence contributes to music-induced analgesia. Pain. 2008 Jan;134(1-2):140-7. doi: 10.1016/j.pain.2007.04.003. Epub 2007 May 25. PMID 17532141